CLINICAL TRIAL: NCT04949646
Title: Intraoperative Neuromonitoring of Pelvic Autonomous Nerve Plexus During Total Mesorectal Excision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Collaborators: General Hospital of Larissa (Other); University of Thessaly (Other)
Responsible Party: Principal Investigator, Perivoliotis Konstantinos, Perivoliotis Konstantinos, Principal Investigator, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PelIONM
Record Dates: First submitted 2021-06-22; First posted 2021-07-02 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Rectal Neoplasms
Keywords: intraoperative; neuromonitoring; pelvic; autonomous; total; mesorectal; excision
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will employ a prospective, parallel randomized-controlled design
Who Masked: Participant
Masking Description: The patient will be blinded regarding the allocation group. Blinding will not exist at the level of the surgeon, the anaesthesiologist, and the investigator responsible for the data recording
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pIONM (Experimental): In the experimental group pIONM will be performed intraoperatively. For the implementation of pIONM, a special device, that allows simultaneous monitoring of sphincter signals and bladder manometry, will be introduced. This device will employ the placement of a bipolar electrode in the internal and external anal sphincter. Moreover, another electrode will be placed on the surrounding tissues. For bladder manometry, the catheter will be connected to the pressure sensor, and subsequently to the pIONM monitor. Intraoperatively, depending on the approach (open or laparoscopic), the respective bipolar stimulator will be used.
  Prior to the initiation of pIONM, urinary bladder will be drained and filled with 200 ml R/L. The pIONM parameters will be the following: 1-25 milliampere current, 30 Hz frequency and 200 μs monophasic pulses.
  Interventions: Other: Pelvic Intraoperative Neuromonitoring
- Control (No Intervention): In the control group pIONM will not be performed intraoperatively

INTERVENTIONS:
Other: Pelvic Intraoperative Neuromonitoring — Pelvic Intraoperative Neuromonitoring (pIONM) allows mapping of the pelvic autonomous plexus during total mesorectal excision (TME).
  Arms: pIONM

SUMMARY:
The purpose of this research protocol is the evaluation of the improvement of the anorectal and urogenital urinary function, alongside the postoperative quality of life after the application of pIONM in patients submitted to TME for rectal cancer.

DETAILED DESCRIPTION:
The introduction of Total Mesorectal Excision (TME) resulted to the improvement of the overall survival and local recurrence rates of rectal cancer patients. However, the associated urogenital and anorectal functional deficit has a significant effect on the postoperative quality of life of the patient. More specifically, the postoperative rates of urogenital and sexual dysfunction that have been reported in the various series, are estimated at the levels of 70% and 90%, respectively. Additionally, TME is associated with the development of the low anterior syndrome (LARS). LARS is characterized by the onset of fecal incontinence, due to injury in the autonomic nerve plexuses that innervate the internal anal sphincter (IAS); who in turn is responsible for the 52-85% anal resting tone. According to a recent study, 38.8% and 33.7% of patients with normal preoperative urogenital function, developed postoperative stool and urine incontinence, respectively.

It becomes apparent that the incidence rates of these complications vary between the various series, mainly due to their small sample size, the lack of comparative data, the short follow up period, the use of non-validated tools and their retrospective design. Several predictive factors of these adverse events have been suggested in the literature, including old age, tumors located less than 12 cm from the anal verge, preoperative radiotherapy and injury to the pelvic autonomous nerves.

The clinical and functional anatomy of the pelvis are quite complex. The inferior hypogastric plexus is formed by the parasympathetic pelvic nerves, deriving from the I2-I4 and the sympathetic hypogastric nerve. It is a neural anatomic structure that carries organ-specific nerve fibers. Visual identification of the plexus is quite difficult, for various reasons, including the complexity of the nerve distribution, the narrow pelvis, the voluminous mesorectum, obesity, previous pelvic operations, neoadjuvant radiotherapy, locally advanced tumors, intraoperative bleeding and the extensive use of diathermy. According to the current literature, identification of the autonomous pelvic plexus is achievable in 72% of cases, whereas partial localization is possible only in 10.7% of patients.

Theoretically, intraoperative neuromonitoring of the pelvic autonomous nerves (pIONM), could quantify intraoperative nerve injuries, while in parallel, contribute to the improvement of the patients' postoperative quality of life. Several pIONM techniques have been described, including intra-urethral and intra-vesical pressure measurements. However, it was found that intermittent neuromonitoring objectifies the macroscopic integrity assessment of the sacral plexus. Recently, a promising technique, based on the simultaneous electromyography of the IAS and bladder manometry was developed, with encouraging results. During pIONM, the surgeon delivers electric stimuli to the autonomic nerve structures through a hand-held stimulator. At the same time, electromyogram changes of the IAS and the external anal sphincter (EAS), alongside intravesical pressure gradients are assessed.

Intraoperative neuromonitoring has been evaluated in several experimental studies. In a recent study, intraoperative simulation of the inferior hypogastric plexus with a bipolar stimulator resulted to the appearance of a measurable and repeatable electromyographic signal from the IAS.

Simultaneous signal processing from the IAS and urinary bladder, improves the, overall, diagnostic accuracy of these techniques. Stabilization of the electrodes outside the surgical field, has been, also, suggested by some researchers. Additionally, experimental studies evaluated the role of pIONM in the minimal invasive TME.

Moreover, the effectiveness of this technique has been a research subject in multiple clinical trials. In another study, where 85 patients underwent TME, after logistic regression, no use of pIONM and neoadjuvant radiotherapy, were identified as independent prognostic factors of postoperative urogenital deficit. Furthermore, the use of pIONM, was associated with a 100% sensitivity and a 96% specificity for the postoperative development of urogenital and anorectal functional complications.

The application of pIONM has been also suggested in the laparoscopic and robotic TME, using specially designed stimulators. In another trial, preservation of the plexus was achieved in 51.7% of patients submitted to a laparoscopic low anterior resection for rectal cancer. During one year follow-up, patients receiving pIONM, displayed a superiority in terms of postoperative urogenital function, as assessed by the IIEF, IPSS and FSFI questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed rectal cancer
* Surgical resection with TME
* <90 years old
* Signed informed consent

Exclusion Criteria:

* Emergency operation
* Presence of pacemaker
* Partial mesorectal excision
* Sepsis or systematic infection
* Physical or mental impairment
* Pregnancy or nursing
* Insufficient preoperative data for the urogenital/ anorectal function
* Lack of compliance with the research process

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-09-19 (Actual); Primary Completion 2027-09-19 (Estimated); Study Completion 2028-09-19 (Estimated)

PRIMARY OUTCOMES:
Change in the quality of life of the patient at 3 months postoperatively, based on the SF-36 questionnaire | Preoperatively, 3 months postoperatively
  Change in the quality of life of the patient, at 3 months postoperatively, compared to the respective preoperative measurements, based on the Short Form 36 (SF-36) questionnaire SF-36: Short Form Survey Minimum Value: 0 Maximum Value: 100 Higher scores indicate a better outcome

SECONDARY OUTCOMES:
Operative time | Intraoperative period
  The total operative time will be recorded. Measurement unit: minutes
Intraoperative bleeding | Intraoperative period
  The total intraoperative blood loss volume will be recorded. Measurement unit: mL
Postoperative discharge time | Maximum time frame 15 days postoperatively
  Postoperative time that the patient can be safely discharged. Measurement unit: hours. The patient will be discharged, when it is ensured that is medically safe to be released. In particular, as the exit time of the patient, will be regarded the time that the patient will fulfil the Clinical Discharge Criteria. More specifically, the patient should meet the following : steady vital signs, be oriented, without nausea or vomiting, mobilized with a steady gait, without a significant bleeding
Postoperative complications | 1 month postoperatively
  Occurrence of postoperative complications (based on Clavien-Dindo classification). If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Negative resection margin | 1 month postoperatively
  Occurrence of negative resection margin. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Local recurrence | 1 year postoperatively
  Occurrence of local recurrence. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Bladder capacity | Preoperatively and 2 months postoperatively
  Urodynamic assessment. Evaluation of bladder capacity. Measurement unit: ml
Bladder compliance | Preoperatively and 2 months postoperatively
  Urodynamic assessment. Evaluation of bladder compliance. Measurement unit: ml/cm H2O
Detrusor pressure at maximum flow | Preoperatively and 2 months postoperatively
  Urodynamic assessment. Evaluation of detrusor pressure at maximum flow. Measurement unit: cm H2O
Maximum urinary flow rate | Preoperatively and 2 months postoperatively
  Urodynamic assessment. Evaluation of maximum urinary flow rate. Measurement unit: ml/s
Voiding volume | Preoperatively and 2 months postoperatively
  Urodynamic assessment. Evaluation of voiding volume. Measurement unit: ml
Post-void residual | Preoperatively and 2 months postoperatively
  Urodynamic assessment. Evaluation of post-void residual. Measurement unit: ml
Anal canal resting phase pressure | Preoperatively and 2 months postoperatively
  High-resolution Anorectal Manometry assessment. Evaluation of anal canal resting phase pressure. Measurement unit: mmHg
Sphincter zone length | Preoperatively and 2 months postoperatively
  High-resolution Anorectal Manometry assessment. Evaluation of sphincter zone length. Measurement unit: cm
Short squeeze test | Preoperatively and 2 months postoperatively
  High-resolution Anorectal Manometry assessment. Evaluation of short squeeze (5sec) pressure. Measurement unit: mmHg
Long squeeze test | Preoperatively and 2 months postoperatively
  High-resolution Anorectal Manometry assessment. Evaluation of long squeeze (30sec) pressure. Measurement unit: mmHg
Cough test | Preoperatively and 2 months postoperatively
  High-resolution Anorectal Manometry assessment. Evaluation of cough test (0 and 50 ml). If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Push test | Preoperatively and 2 months postoperatively
  High-resolution Anorectal Manometry assessment. Evaluation of push test (0 and 50 ml). If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
RAIR test | Preoperatively and 2 months postoperatively
  High-resolution Anorectal Manometry assessment. Evaluation of rectoanal inhibitory reflex (RAIR) test (20 and 50 ml). If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Difference in the quality of life of the patient, based on the SF-36 questionnaire | Preoperatively, 6, 12, 24 months postoperatively
  Difference in the quality of life of the patient, at 6, 12, 24 months postoperatively, compared to the respective preoperative measurements, based on the Short Form 36 (SF-36) questionnaire SF-36: Short Form Survey Minimum Value: 0 Maximum Value: 100 Higher scores indicate a better outcome
Difference in the erectile function of the patient, based on the IIEF questionnaire | Preoperatively, 3, 6, 12, 24 months postoperatively
  Difference in the erectile function of the patient, at 3, 6, 12, 24 months postoperatively, compared to the respective preoperative measurements, based on the International Index of Erectile Function (IIEF) questionnaire IIEF: International Index of Erectile Function Minimum Value: 0 Maximum Value: 5 Higher scores indicate a better outcome
Difference in the sexual function of the patient, based on the FSFI questionnaire | Preoperatively, 3, 6, 12, 24 months postoperatively
  Difference in the sexual function of the patient, at 3, 6, 12, 24 months postoperatively, compared to the respective preoperative measurements, based on the Female Sexual Function Index (FSFI) questionnaire FSFI: Female Sexual Function Index Minimum Value: 2 Maximum Value: 36 Higher scores indicate a better outcome
Difference in the prostate symptoms of the patient, based on the IPSS questionnaire | Preoperatively, 3, 6, 12, 24 months postoperatively
  Difference in the prostate symptoms of the patient, at 3, 6, 12, 24 months postoperatively, compared to the respective preoperative measurements, based on the International Prostate Symptom Score (IPSS) questionnaire IPSS: International Prostate Symptom Score Minimum Value: 0 Maximum Value: 35 Higher scores indicate a worse outcome
Difference in the low anterior syndrome symptoms of the patient, based on the LARS questionnaire | Preoperatively, 3, 6, 12, 24 months postoperatively
  Difference in the low anterior syndrome symptoms of the patient, at 3, 6, 12, 24 months postoperatively, compared to the respective preoperative measurements, based on the Low Anterior Resection Syndrome (LARS) questionnaire LARS: Low Anterior Resection Syndrome Minimum Value: 0 Maximum Value: 42 Higher scores indicate a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Tepetes, Prof, Study Director — Department of Surgery, University Hospital of Larissa; Konstantinos Perivoliotis, MD, Principal Investigator — Department of Surgery, University Hospital of Larissa
Locations (1):
- University Hospital of Larissa, Larissa, Greece

IPD SHARING:
Plan to Share IPD: No
No plan to share individual patient data

REFERENCES:
- [Background] Kauff DW, Kempski O, Koch KP, Huppert S, Hoffmann KP, Lang H, Kneist W. Continuous intraoperative monitoring of autonomic nerves during low anterior rectal resection: an innovative approach for observation of functional nerve integrity in pelvic surgery. Langenbecks Arch Surg. 2012 Jun;397(5):787-92. doi: 10.1007/s00423-011-0900-x. Epub 2012 Feb 15. PMID 22350611
- [Background] Kauff DW, Lang H, Kneist W. Risk Factor Analysis for Newly Developed Urogenital Dysfunction after Total Mesorectal Excision and Impact of Pelvic Intraoperative Neuromonitoring-a Prospective 2-Year Follow-Up Study. J Gastrointest Surg. 2017 Jun;21(6):1038-1047. doi: 10.1007/s11605-017-3409-y. Epub 2017 Apr 4. PMID 28378317
- [Background] Wallner C, Lange MM, Bonsing BA, Maas CP, Wallace CN, Dabhoiwala NF, Rutten HJ, Lamers WH, Deruiter MC, van de Velde CJ; Cooperative Clinical Investigators of the Dutch Total Mesorectal Excision Trial. Causes of fecal and urinary incontinence after total mesorectal excision for rectal cancer based on cadaveric surgery: a study from the Cooperative Clinical Investigators of the Dutch total mesorectal excision trial. J Clin Oncol. 2008 Sep 20;26(27):4466-72. doi: 10.1200/JCO.2008.17.3062. PMID 18802159
- [Background] Kauff DW, Kronfeld K, Gorbulev S, Wachtlin D, Lang H, Kneist W. Continuous intraoperative monitoring of pelvic autonomic nerves during TME to prevent urogenital and anorectal dysfunction in rectal cancer patients (NEUROS): a randomized controlled trial. BMC Cancer. 2016 May 21;16:323. doi: 10.1186/s12885-016-2348-4. PMID 27209237
- [Background] Delacroix SE Jr, Winters JC. Voiding dysfunction after pelvic colorectal surgery. Clin Colon Rectal Surg. 2010 Jun;23(2):119-27. doi: 10.1055/s-0030-1254299. PMID 21629630
- [Background] Kneist W, Kauff DW, Rahimi Nedjat RK, Rink AD, Heimann A, Somerlik K, Koch KP, Doerge T, Lang H. Intraoperative pelvic nerve stimulation performed under continuous electromyography of the internal anal sphincter. Int J Colorectal Dis. 2010 Nov;25(11):1325-31. doi: 10.1007/s00384-010-1015-5. Epub 2010 Jul 27. PMID 20661601
- [Background] Moszkowski T, Kauff DW, Wegner C, Ruff R, Somerlik-Fuchs KH, Kruger TB, Augustyniak P, Hoffmann KP, Kneist W. Extracorporeal Stimulation of Sacral Nerve Roots for Observation of Pelvic Autonomic Nerve Integrity: Description of a Novel Methodological Setup. IEEE Trans Biomed Eng. 2018 Mar;65(3):550-555. doi: 10.1109/TBME.2017.2703951. Epub 2017 May 12. PMID 28504930
- [Background] Kauff DW, Koch KP, Somerlik KH, Heimann A, Hoffmann KP, Lang H, Kneist W. Online signal processing of internal anal sphincter activity during pelvic autonomic nerve stimulation: a new method to improve the reliability of intra-operative neuromonitoring signals. Colorectal Dis. 2011 Dec;13(12):1422-7. doi: 10.1111/j.1463-1318.2010.02510.x. PMID 21087387
- [Background] Kauff DW, Moszkowski T, Wegner C, Heimann A, Hoffmann KP, Kruger TB, Lang H, Kneist W. Transcutaneous sacral nerve stimulation for intraoperative verification of internal anal sphincter innervation. Neurogastroenterol Motil. 2017 Dec;29(12). doi: 10.1111/nmo.13140. Epub 2017 Jul 6. PMID 28681496
- [Background] Schiemer JF, Juo YY, Sanaiha Y, Lin AY, Kazanjian K, Lang H, Kneist W. Application of a newly designed microfork probe for robotic-guided pelvic intraoperative neuromapping. J Minim Access Surg. 2019 Apr-Jun;15(2):182-183. doi: 10.4103/jmas.JMAS_12_18. PMID 29582794
- [Background] Kauff DW, Koch KP, Somerlik KH, Hoffmann KP, Lang H, Kneist W. Evaluation of two-dimensional intraoperative neuromonitoring for predicting urinary and anorectal function after rectal cancer surgery. Int J Colorectal Dis. 2013 May;28(5):659-64. doi: 10.1007/s00384-013-1662-4. Epub 2013 Feb 26. PMID 23440364
- [Background] Grade M, Beham AW, Schuler P, Kneist W, Ghadimi BM. Pelvic intraoperative neuromonitoring during robotic-assisted low anterior resection for rectal cancer. J Robot Surg. 2016 Jun;10(2):157-60. doi: 10.1007/s11701-015-0556-6. Epub 2015 Dec 24. PMID 26705113
- [Background] Kneist W, Kauff DW, Naumann G, Lang H. Resection rectopexy--laparoscopic neuromapping reveals neurogenic pathways to the lower segment of the rectum: preliminary results. Langenbecks Arch Surg. 2013 Apr;398(4):565-70. doi: 10.1007/s00423-013-1064-7. Epub 2013 Feb 23. PMID 23435617
- [Background] Schiemer JF, Zimniak L, Hadzijusufovic E, Lang H, Kneist W. Novel multi-image view for neuromapping meets the needs of the robotic surgeon. Tech Coloproctol. 2018 Jun;22(6):445-448. doi: 10.1007/s10151-018-1804-3. Epub 2018 Jun 4. PMID 29868993
- [Background] Zhou MW, Huang XY, Chen ZY, Li ZY, Zhou YM, Yang Y, Wang ZH, Xiang JB, Gu XD. Intraoperative monitoring of pelvic autonomic nerves during laparoscopic low anterior resection of rectal cancer. Cancer Manag Res. 2018 Dec 31;11:411-417. doi: 10.2147/CMAR.S182181. eCollection 2019. PMID 30643466
- [Background] Fang JF, Wei B, Zheng ZH, Chen TF, Huang Y, Huang JL, Lei PR, Wei HB. Effect of intra-operative autonomic nerve stimulation on pelvic nerve preservation during radical laparoscopic proctectomy. Colorectal Dis. 2015 Dec;17(12):O268-76. doi: 10.1111/codi.13115. PMID 26362914
- [Background] Kneist W, Junginger T. Validity of pelvic autonomic nerve stimulation with intraoperative monitoring of bladder function following total mesorectal excision for rectal cancer. Dis Colon Rectum. 2005 Feb;48(2):262-9. doi: 10.1007/s10350-004-0797-3. PMID 15714244
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Rosier PFWM, Schaefer W, Lose G, Goldman HB, Guralnick M, Eustice S, Dickinson T, Hashim H. International Continence Society Good Urodynamic Practices and Terms 2016: Urodynamics, uroflowmetry, cystometry, and pressure-flow study. Neurourol Urodyn. 2017 Jun;36(5):1243-1260. doi: 10.1002/nau.23124. Epub 2016 Dec 5. PMID 27917521
- [Background] Pappa E, Kontodimopoulos N, Niakas D. Validating and norming of the Greek SF-36 Health Survey. Qual Life Res. 2005 Jun;14(5):1433-8. doi: 10.1007/s11136-004-6014-y. PMID 16047519
- [Background] Rosen RC, Riley A, Wagner G, Osterloh IH, Kirkpatrick J, Mishra A. The international index of erectile function (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology. 1997 Jun;49(6):822-30. doi: 10.1016/s0090-4295(97)00238-0. PMID 9187685
- [Background] Mourikis I, Antoniou M, Matsouka E, Vousoura E, Tzavara C, Ekizoglou C, Papadimitriou GN, Vaidakis N, Zervas IM. Anxiety and depression among Greek men with primary erectile dysfunction and premature ejaculation. Ann Gen Psychiatry. 2015 Oct 29;14:34. doi: 10.1186/s12991-015-0074-y. eCollection 2015. PMID 26516337
- [Background] Stephenson KR, Toorabally N, Lyons L, M Meston C. Further Validation of the Female Sexual Function Index: Specificity and Associations With Clinical Interview Data. J Sex Marital Ther. 2016 Jul 3;42(5):448-61. doi: 10.1080/0092623X.2015.1061078. Epub 2015 Jun 22. PMID 26098130
- [Background] Zachariou A, Filiponi M, Kirana PS. Translation and validation of the Greek version of the female sexual function index questionnaire. Int J Impot Res. 2017 Jul;29(4):171-174. doi: 10.1038/ijir.2017.18. Epub 2017 Apr 20. PMID 28424501
- [Background] Bayoud Y, de la Taille A, Ouzzane A, Ploussard G, Allory Y, Yiou R, Vordos D, Hoznek A, Salomon L. International Prostate Symptom Score is a predictive factor of lower urinary tract symptoms after radical prostatectomy. Int J Urol. 2015 Mar;22(3):283-7. doi: 10.1111/iju.12681. Epub 2015 Jan 22. PMID 25612145
- [Background] Konstantinidis C, Samarinas M, Andreadakis S, Xanthis S, Skriapas K. Lower urinary tract symptoms associated with benign prostatic hyperplasia: combined treatment with fesoterodine fumarate extended-release and tamsulosin--a prospective study. Urol Int. 2013;90(2):156-60. doi: 10.1159/000345050. Epub 2012 Dec 5. PMID 23221480
- [Background] Juul T, Ahlberg M, Biondo S, Emmertsen KJ, Espin E, Jimenez LM, Matzel KE, Palmer G, Sauermann A, Trenti L, Zhang W, Laurberg S, Christensen P. International validation of the low anterior resection syndrome score. Ann Surg. 2014 Apr;259(4):728-34. doi: 10.1097/SLA.0b013e31828fac0b. PMID 23598379
- [Background] Liapi A, Mavrantonis C, Lazaridis P, Kourkouni E, Zevlas A, Zografos G, Theodoropoulos G. Validation and comparative assessment of low anterior resection syndrome questionnaires in Greek rectal cancer patients. Ann Gastroenterol. 2019 Mar-Apr;32(2):185-192. doi: 10.20524/aog.2019.0350. Epub 2019 Jan 15. PMID 30837792
- [Background] O'Leary DP, Fide CJ, Foy C, Lucarotti ME. Quality of life after low anterior resection with total mesorectal excision and temporary loop ileostomy for rectal carcinoma. Br J Surg. 2001 Sep;88(9):1216-20. doi: 10.1046/j.0007-1323.2001.01862.x. PMID 11531870
- [Background] MERCURY Study Group. Diagnostic accuracy of preoperative magnetic resonance imaging in predicting curative resection of rectal cancer: prospective observational study. BMJ. 2006 Oct 14;333(7572):779. doi: 10.1136/bmj.38937.646400.55. Epub 2006 Sep 19. PMID 16984925
- [Background] Carrington EV, Heinrich H, Knowles CH, Fox M, Rao S, Altomare DF, Bharucha AE, Burgell R, Chey WD, Chiarioni G, Dinning P, Emmanuel A, Farouk R, Felt-Bersma RJF, Jung KW, Lembo A, Malcolm A, Mittal RK, Mion F, Myung SJ, O'Connell PR, Pehl C, Remes-Troche JM, Reveille RM, Vaizey CJ, Vitton V, Whitehead WE, Wong RK, Scott SM; All members of the International Anorectal Physiology Working Group. The international anorectal physiology working group (IAPWG) recommendations: Standardized testing protocol and the London classification for disorders of anorectal function. Neurogastroenterol Motil. 2020 Jan;32(1):e13679. doi: 10.1111/nmo.13679. Epub 2019 Aug 12. PMID 31407463
- [Background] Chung F, Chan VW, Ong D. A post-anesthetic discharge scoring system for home readiness after ambulatory surgery. J Clin Anesth. 1995 Sep;7(6):500-6. doi: 10.1016/0952-8180(95)00130-a. PMID 8534468
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190

DOCUMENTS (2):
  • Study Protocol (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT04949646/Prot_000.pdf
  • Informed Consent Form (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT04949646/ICF_001.pdf